CLINICAL TRIAL: NCT03832192
Title: Care.Coach Avatars for Improvement of Outcomes in Hospitalized Elders, Including Mitigation of Falls and Delirium, Through Psychosocial Support and Protocol-Driven Interventions Based on the Hospital Elder Life Program: a Multi-Site Clinical Study
Brief Title: Care.Coach Avatars for Improvement of Outcomes in Hospitalized Elders, Including Mitigation of Falls and Delirium: a Multi-Site Clinical Study
Acronym: AvatarHELP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Victor Wang (Industry)
Collaborators: National Institute of Nursing Research (NINR) (NIH); Pace University (Other)
Responsible Party: Sponsor-Investigator, Victor Wang, Principal Investigator, care.coach corporation
Organization: care.coach corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1R44NR017842-02 (NIH)
Record Dates: First submitted 2019-01-29; First posted 2019-02-06 (Actual); Results first posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-07

CONDITIONS: Delirium; Fall Injury
Keywords: patient satisfaction; HCAHPS; loneliness; delirium; falls; HELP; hospitals; geriatrics; elder care
MeSH Terms: conditions — Delirium; Patient Satisfaction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- care.coach Avatar (Experimental)
  Interventions: Behavioral: care.coach Avatar (HELP-Protocolized)
- Control (No Intervention)

INTERVENTIONS:
Behavioral: care.coach Avatar (HELP-Protocolized) — care.coach human-in-the-loop avatar system with software-directed protocols based on the Hospital Elder Life Program (HELP).
  Arms: care.coach Avatar

SUMMARY:
Through NINR project 1R44NR017842-01 which preceded the present study, the investigators enhanced the care.coach avatar platform to incorporate a robust suite of evidence-based protocols based on the Hospital Elder Life Program (HELP), and to leverage an integration with hospital-based electronic medical record (EMR) systems. In the present study, the investigators seek to validate the efficacy of the new avatar platform, as measured by reduction in falls, delirium, and patient sitter utilization. Also, the investigators seek to gather patient and outcomes data at a scale sufficient to begin developing machine learning algorithms for intelligent, automatic assignment of protocols to maximize patient engagement and clinical efficacy, and for intelligent, automatic screening of delirium to assist care teams in positive identification of delirium. Therefore, the present study comprises a two-year randomized between-groups comparison across multiple hospitals to compare outcomes with the new generation of care.coach avatars as the intervention versus usual care only as the control. Each study group will be geographically distributed across participating research sites: initially MediSys Health Network's Jamaica Hospital Medical Center in New York, with additional hospitals to join the study over the course of two years.

ELIGIBILITY:
Inclusion Criteria:

* fall/delirium risk (may be based purely on age at the election of each site, e.g. 65+)

Exclusion Criteria:

* aggression or combativeness with intent to harm self or others
* severe hearing impairment and simultaneous severe vision impairment, despite assistive devices
* no comprehension of either Spanish or English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2021-01-07 (Actual); Study Completion 2021-01-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Jamaica Hospital Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: care.coach human-in-the-loop avatars for psychosocial support, health coaching, and care coordination — http://care.coach

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: HELP-protocolized digital avatar with daily nurse student check-in
- Control: Usual care with daily nurse student social check-in
Period: Overall Study
Arm/Group | Intervention | Control
Started | 152 | 149
Completed | 0 | 0
Not Completed | 152 | 149
Not completed — Participants are disenrolled upon hospital discharge. | 152 | 149

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 152 | 149 | 301
Age, Continuous [Mean (Standard Deviation); unit: years] | 76 (9) | 75 (8) | 76 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 58 | 134
  Male | 76 | 91 | 167
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 26 | 52
  Not Hispanic or Latino | 119 | 117 | 236
  Unknown or Not Reported | 7 | 6 | 13
Short Portable Mental Status Questionnaire [Mean (Standard Deviation); unit: number of questions incorrectly answered] — 0 to 10 questions incorrectly answered; greater number indicates worse cognitive performance
  number of questions incorrectly answered | 2.0 (1.8) | 2.6 (2.4) | 2.3 (2.1)
Confusion Assessment Method [Number; unit: number of positive screens] — Delirium screening algorithm resulting in either positive of negative presence of delirium
  number of positive screens | 23 | 8 | 31
Memorial Delirium Assessment Scale [Mean (Standard Deviation); unit: scores on a scale] — 10 severity items rated 0 to 3 points for a maximum total score of 30 points, with higher scores representing more severe delirium
  scores on a scale | 8.2 (4.6) | 14.3 (4.6) | 12.6 (5.3)

OUTCOME MEASURES:

1. Primary Outcome: Incident Delirium Rate
Description: For each patient without prevalent delirium (each patient who screens negative per the Confusion Assessment Method [CAM] upon study enrollment, which is assumed to be within 24 hours of admission to the hospital unit), Incident Delirium is indicated by any positive CAM screen during the patient's study enrollment period, with CAM screens being performed at least daily (the final CAM screen is assumed to be within 24 hours of discharge from the hospital unit). Incident Delirium is thus a binary variable (true/false) for each patient, and the rate of Incident Delirium will be compared across study groups, with a lower rate being desirable.
Time Frame: From beginning to end of each participant's inpatient stay, an average of 4 days
Population: Patients without prevalent delirium and have a final CAM screen on record
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 87 | 65
Participants | 6 | 0

2. Secondary Outcome: Delirium Resolution Rate
Description: For each patient with prevalent delirium (each patient who screens positive per the Confusion Assessment Method [CAM] upon study enrollment, which is assumed to be within 24 hours of admission to the hospital unit), delirium will be considered resolved if the patient's final CAM screen (which is assumed to be within 24 hours prior to discharge from the hospital unit) indicates no delirium. Delirium Resolution is thus a binary variable (true/false) for each patient, and the rate of successful Delirium Resolution will be compared across study groups, with a higher rate being desirable.
Time Frame: From beginning to end of each participant's inpatient stay, an average of 4 days
Population: Patients with prevalent delirium and a final CAM screen on record
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 5 | 8
Participants | 3 | 5

3. Secondary Outcome: Change in Cognitive Function
Description: For each patient, the Short Portable Mental Status Questionnaire (SPMSQ) is administered to measure cognitive function (0-10 errors, more errors indicating greater cognitive impairment) upon enrollment and upon dis-enrollment from the study. Change in Cognitive Function is the difference from the enrollment SPMSQ score to the dis-enrollment SPMSQ score. Change in Cognitive Function will be compared across study groups, with a larger numerical reduction being desirable.
Time Frame: From beginning to end of each participant's inpatient stay, an average of 4 days
Population: Patients with both pre- and post-test data on record
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 87 | 68
score on a scale | 0.14 (1.8) | -0.15 (2.4)

4. Other Pre Specified Outcome: Change in Delirium Severity
Description: For each patient screened delirium positive on the Confusion Assessment Method (CAM), the Memorial Delirium Assessment Scale (MDAS) is administered to measure delirium severity upon enrollment and upon dis-enrollment from the study. Change in Delirium Severity is the difference from the enrollment MDAS score to the dis-enrollment MDAS score. Change in Delirium Severity will be compared across study groups, with a larger numerical reduction being desirable.
Time Frame: From beginning to end of each participant's inpatient stay, an average of 4 days
Population: Patients with both pre- and post-test MDAS data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 1 | 1
score on a scale | -2 | -5

ADVERSE EVENTS:
Time Frame: From beginning to end of each participant's inpatient stay, an average of 4 days
Description: The usual definition of a "serious adverse event" includes an inpatient hospitalization, but all subjects are already hospitalized and therefore we are focusing on deaths unless there is a usually-defined serious or non-serious adverse event that is considered attributable to study participation.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/152 | 0/149
Serious Adverse Events (participants affected / at risk) | 0/152 | 0/149
Other Adverse Events (participants affected / at risk) | 0/152 | 0/149

LIMITATIONS AND CAVEATS:
Fall & patient sitter data were not recorded at the first site. Secondary sites that were to record such data were stalled by COVID. Post-tests were missing for many patients, due largely to hospital discharges occurring before researchers could conduct post-tests. Incident delirium cases were too few to draw conclusions (far below the rate suggested by literature). The team began to mitigate these data integrity problems, but were not able to rebuild a viable research assistant team post-COVID.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-28): https://cdn.clinicaltrials.gov/large-docs/92/NCT03832192/Prot_SAP_000.pdf